CLINICAL TRIAL: NCT07091786
Title: Complete Digital Workflow for Construction of Full Arch Implant Supported Screw Retained Restoration: Clinical Evaluation of Titanium-zirconium Versus Peek-composite
Brief Title: Complete Digital Workflow
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: J0204023RP
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Digital Intervention
MeSH Terms: interventions — Dental Prosthesis, Implant-Supported

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group1 (Active Comparator): • the titanium group involved patients who will be received ISFCDs with individual zirconium veneers
  Interventions: Device: Implant supported prosthesis
- group 2 (Active Comparator): The PEEK group included patients who will be received ISFCDs with individual PMMA composite veneers cemented onto a CAD-CAM PEEK framework
  Interventions: Device: Implant supported prosthesis

INTERVENTIONS:
Device: Implant supported prosthesis — implant supported full arch prosthesis

SUMMARY:
This study will aim to clinical evaluation of titanium-zirconium and peek-composite of screw retained prosthesis used for rehabilitation of edentulous patients using Complete digital workflow for construction of full arch implant supported screw retained restoration.

ELIGIBILITY:
Inclusion Criteria:

* i- Edentulous jaws ii- Good oral hygiene and good compliance. iii- Angel's class I maxillo-mandibular relationship and a minimum of 16mm mandibular restorative space at the estimated occlusal vertical dimension. This will be verified by recoding a tentative jaw relation iv- Adequate bone height and width for placement of standard diameter implants. A cone beam computerized tomographic scan will be taken prior to surgery to determine the bone quality and bone volume

Exclusion Criteria:i- Systemic disease: uncontrolled diabetes mellitus, cardiovascular disease, immunodeficiency disorders, blood disorders such as coagulation disorders, severe osteoporosis, and any metabolic disease that might influence the rate of bone resorption ii- Long-term medication use: steroid, anti-epileptic drugs, drugs favoring gingival overgrowth, bispho- sphonates (bisphosphonate injections or more than 4 years of oral bisphosphonate use), and any medi- cation that influences the rate of bone loss or sur- vival of dental implants. iii- Infection of human immunodeficiency virus, hepatitis B virus, or syphilis iv- Bruxism v- Maxillofacial tumor

-

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Prosthetic complication | one year
  Complication will be evaluated clinically
Marginal Bone loss | one year
  Bone loss will be evaluated Radiographically around dental implants

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No